CLINICAL TRIAL: NCT02641769
Title: Intra-Testicular Transplantation of Purified Autologous Clusters of Differentiation (CD) 34+,133+, and Mesenchymal Stem Cells for Treatment of Non-Obstructive Azoospermia Male Infertility.
Brief Title: Intra-Testicular Transplantation of Autologous Stem Cells for Treatment of Non-Obstructive Azoospermia Male Infertility.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-INF1
Record Dates: First submitted 2015-12-07; First posted 2015-12-29 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Non-obstructive Azoospermia
MeSH Terms: interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell Transplantation (Other): intervention with transplantation of autologous purified stem cells
  Interventions: Biological: Stem Cell Transplantation

INTERVENTIONS:
Biological: Stem Cell Transplantation — intervention with transplantation of autologous purified stem cells

SUMMARY:
This is an open label, single arm, single center investigation to assess the safety and efficacy of purified adult autologous bone marrow derived CD34+, CD133+, and mesenchymal stem cells injected into the seminiferous tubules and testis, through a 12 week follow-up period. The investigators' selected model of research is based on maximizing the efficiency of the approach by choosing an autologous pattern which preserves the genetic make-up of an individual that is vital in infertility conditions. Additionally the approach involves injecting a combination of different but purified cell types which all aid in the retrieval of spermatogenesis, and the generation of mature spermatozoa. Expected outcomes of this study are defined in general improvements in infertile patients in regards of testicular morphology, sexual function, semen quality, development of primary or secondary spermatocytes, spermatids, or mature spermatozoa in the testis, seminiferous tubules, or semen.

DETAILED DESCRIPTION:
Non-obstructive azoospermia (NOA) is generally considered a non-medically manageable cause of male infertility. These patients, who constitute up to 10% of all infertile men, have abnormal spermatogenesis as the cause of their azoospermia. The etiology affecting approximately 60% of azoospermic men, includes non-obstructive causes of azoospermia, including toxic exposures or abnormal testicular development. NOA results from either primary testicular failure (elevated Luteinizing Hormone (LH), Follicle stimulating hormone (FSH), small testes affecting up to 10% of men presenting with infertility), secondary testicular failure (congenital hypogonadotropic hypogonadism with decreased LH and FSH, small testes), or incomplete or ambiguous testicular failure (either increased FSH and normal volume testes, normal FSH and small testes, or normal FSH and normal testis volume). Prior to microsurgical testicular sperm retrieval techniques and IVF/ICSI, donor insemination was the only option available to men with NOA. The establishment of in vitro fertilization using intracytoplasmic sperm injection (ICSI) as a standard treatment modality has resulted in a number of these men successfully fathering a child through surgically retrieved sperm from the testis. The challenge, however, is to improve their spermatogenic function to enable the appearance of sperm in their ejaculate or to improve the chances of a successful retrieval from the testis for ICSI.

The initial evaluation aims at resolving the following issues: (1) confirming azoospermia, (2) differentiating obstructive from non-obstructive etiology, (3) assessing for the presence of reversible factors and (4) evaluating for the presence of genetic abnormalities. An elevated follicle-stimulating hormone (FSH) level or an absence of normal spermatogenesis by testicular histology in the presence of azoospermia is generally considered sufficient evidence of a non-obstructive etiology. The most common reversible factors that need to be ruled out include recent exogenous hormone administration, severe febrile illnesses, chemotherapy/radiation or prolonged antibiotic use.

During past few years a considerable progress in the derivation of male germ cells from pluripotent stem cells has been made. These studies provide a desirable experimental model for elucidating underlying molecular mechanism of male germ cell development and potential strategies for producing haploid germ cells for the treatment of male infertility. Spermatogenesis is a complex process by which spermatogonial stem cells (SSC) self-renew and differentiate into haploid spermatozoa. In mammals, this process takes place in the seminiferous tubules of testis, which provide a functional niche for male germ cells and involve three major stages: mitosis, meiosis, and spermiogenesis. Errors at any stage of spermatogenesis can result in subfertility and infertility.

Researchers are currently developing alternative treatment options for these men involving stem cells. It has been verified that mouse induced pluripotent stem cells (iPSCs) can form functional spermatozoa. Functional assays have shown that spermatozoa generated from iPSCs were capable of fertilizing the oocytes after intracytoplasmatic injection and giving rise to fertile offspring following embryo transfer. So far, functional male gametes from human iPSCs have not been obtained.

There are two possible approaches in generating of male germ cells from pluripotent stem cells: in vitro differentiation into advanced, haploid cell products or combined in vitro differentiation and in vivo transplantation. However, the originality of this study is illustrated in the transplantation of purified autologous CD34+/CD133+ and mesenchymal bone marrow stem cells (BMSCs) into infertile patients without in vitro breeding, culture, or manipulation thus avoiding in vitro cell propagation risks as genetic mutations and DNA changes. The cells are withdrawn and injected back into the patient on the very same day of the procedure, hence conferring the highest safety and efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

* Infertile males with confirmed diagnosis of non-obstructive azoospermia (NOA)

Exclusion Criteria:

* Patients with Obstructive Azoospermia (OA)
* Previous surgical history in Testis
* Patients with infectious genital diseases
* Patients with anatomical abnormalities of the genital tract
* Patients with major medical problems as malignancies
* Chromosomal aberration (e.g. Y microdeletion, trisomy….)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-06 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Appearance of different germ cells in testicles through the progress of spermatogenesis will be assessed by the count of cells using histological studies. | 12 months

SECONDARY OUTCOMES:
General improvements of testicular morphology will be assessed with histological studies. | 12 months
Improvement in sexual function will be assessed using a questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adeeb AlZoubi, PhD, Principal Investigator — Stem Cells of Arabia
Locations (1):
- Stem Cells of Arabia, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided